CLINICAL TRIAL: NCT04949672
Title: Pathology Assessment of Mesorectal Fascia and Specimen Quality After TME by Laparoscopic, Open, TransAnal and Robotic Approaches (LOTARTME)
Brief Title: Pathology Assessment of Mesorectal Fascia After TME by Laparoscopic, Open, TransAnal and Robotic Approaches (LOTARTME)
Acronym: LOTARTME
Status: Completed | Type: Observational
Sponsor: San Giovanni Addolorata Hospital (Other)
Responsible Party: Principal Investigator, Marco Maria Lirici, Professor of Surgery, San Giovanni Addolorata Hospital
Other Study IDs: SGAddolorataH
Record Dates: First submitted 2021-06-02; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Rectal Cancer; Surgery
Keywords: TME; TransAnal TME; Mesorectal Fascia; Rectal Cancer Surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Open TME: Total Mesorectal Excision (TME) is the gold standard surgical treatment of rectal cancer. According to the technique first described by Bill Heald, TME entails the resection of the rectum including the whole mesorectal fat and an intact mesorectal fascia. Open TME is accomplished through a midline xifo-umbilical laparotomy and requires a complete mobilization of the left colon and central ligature of inferior mesenteric artery and vein.
- Laparoscopic TME: Laparoscopic TME mirrors the procedure performed through laparotomy with the same operative steps and performing rectal resection including the excision of the surrounding mesorectal fat and fascia.
- Robotic TME: Robotic TME mirrors the procedure described by Bill Heald for open surgery but the operation is performed by the master-slave DaVinci System under 3D laparoscopic guidance. The rectal resection is performed including mesorectal fat and fascia.
- TransAnal TME: TaTME has first described by Antonio Lacy in 2012. This procedure has two steps: abdominal and perineal. The abdominal step is performed through a laparoscopic approach as described for laparoscopic TME but the caudal dissection is stopped right below the level of the peritoneal rectal reflection (Douglas pouch). The perineal step is accomplished transanally inserting a specially designed platform into the anal canal and performing the total mesorectal excision under endoscopic guidance.

SUMMARY:
TME is the gold standard surgical treatment of rectal cancer. Specimen quality, integrity of mesorectal fascia and lymph nodes harvest are expression of radicality and good surgery. The LOTARTME study is designed to assess which of the open, laparoscopic, robotic and endoscopic transanal approach is superior. Primary outcome is the evaluation of completeness of mesorectal fascia according to Quirke classification. Secondary outcomes are lymph nodes harvest, local recurrences, overall survivals, cancer related survivals. Inclusion criteria: any patient of any age and sex undergoing to intent-to-treat surgery operated by experienced surgeon. Exclusion criteria: patients with rectal cancer undergoing palliative surgery or multivisceral resection; all patients operated by less experienced surgeons. Study period January 1, 2017 - June 30 2021 and patients enrollment: January 1, 2017 - December 31, 2020. Data collection and analysis: data are collected in a prospective database and statical analysis is carried out using AnalystSoft StatPlus for Windows Software.

DETAILED DESCRIPTION:
Developed in 1992 by Heald Total Mesorectal Excision improved the long-term results of rectal cancer treatment with overall survivals increasing up to 80% and local recurrences decreasing down to 4%. Notwithstanding the introduction of laparoscopy and robotic technology and their application in the field of rectal cancer surgery in the last decades, no further improvement of rectal cancer survivals have been reported. Actually, completeness of mesorectal fat and fascia excision seems not to be improved with these new approaches, compared to standard open surgery. It has been proved that local recurrences are strictly related to the quality of TME and are significantly higher when mesorectal fascia is incomplete according to Quirke classification. In 2012 A. Lacy first reported the transanal approach to TME, developed to overcome the high challenges represented by low rectal dissection when difficult anatomy is present (i.e. obese pts, narrow pelvis, bulging tumors) that may impair the quality of surgical specimen and, therefore, increase the incidence of local recurrences and, indirectly, overall cancer related survivals. There is an ongoing clinical trial (COLOR III) that has been designed to assess whether long term results after TaTME are similar, better or worse than those of open or laparoscopic TME. Until then scientists and researchers may evaluate the effectiveness of TaTME compared to other surgical approaches (open, laparoscopic, robotic) assessing the quality of surgical specimens (i.e. completeness of mesorectal excision and integrity of mesorectal fascia according to Quirke classification). Investigators have designed a prospective observational cohort study assessing the quality of specimen and mesorectal fascia in all patients undergoing TME through an open, laparoscopic, robotic and transanal (TaTME) approach between January 2017 and December 2020. All patients have been followed-up with a required minimum follow-up of 6 months. Therefore, the study was terminated on June 2021. Inclusion criteria were: any patient of any age and sex undergoing intent-to-treat surgery operated by experienced surgeon (with ≥ 100 TME performed). Exclusion criteria: patients with rectal cancer undergoing palliative surgery or multivisceral resection, all patients operated by less experienced surgeons (< 100 TME performed).

Objective of the study:

Assessing the quality of the specimen after TME carried out through laparoscopic, open, robotic and endoscopic transanal approach; evaluating whether TaTME might be superior the other approaches in term of radicality of surgery and local recurrencies.

Primary outcome:

Quirke classification of mesorectal fat and fascia completeness. Three grade classification: complete, nearly complete, incomplete.

Secondary outcomes Lymph node harvest Local recurrences Overall survivals Cancer specific survivals Pathology assessment

A fresh specimen or in vacuum packing is sent for macroscopic assessment to the pathologist. The specimen is dealt as follows:

1) assessment of mesorectum quality; 2) ink painting of specimen non-peritonealized bare areas 3) the specimen is opened along the anterior aspect from the top and the bottom, leaving the bowel intact at a level just above and just below the tumour; 4) placement of formalin-soaked gauze wicks into the unopened ends of the bowel; 5) the specimen is fixed in 10% buffered formalin for at least 48 hours.

The fixed specimen is dealt as follows:

1) 3-5 mm intervals slices through the unopened rectum; 2) slices inspection to note: extent of tumour and the closest distance of tumour to the Circumferential Resection Margin (CRM); positive nodes and the distance of any positive node to the CRM; anterior, posterior or lateral closest distance of tumour to CRM; 3) lymph nodes detection within the fat away from the tumour

Block selection according to the followings:

1) tumor blocks showing closest CRM; 2) tumor blocks showing luminal aspect, 3) all lymph nodes; 4) any polyps; 5) proximal and distal resection margins (distal margin includes both mucosa and mesorectum).

The pathologist examined the specimen in a blinded fashion (unaware of the name of the operating surgeon and the technique performed).

Data are collected in a prospective database. Statistical analysis is carried out with AnalystSoft StatPlus for Windows Software. Chi-square test and chi-square test with Yates correction are used considering p-value significative at p<.05.

ELIGIBILITY:
Inclusion Criteria:

* intent to treat procedures
* procedures performed by experienced surgeons (minimum of 100 TME)

Exclusion Criteria:

* palliation surgery
* multivisceral resections
* procedures performed by inexperienced surgeons (less of 100 TME)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stage 1 and 2 rectal cancer patients (preoperative assessment) undergoing surgery without neoadjuvant chemoradiation therapy.
  Stage 3 and 4 rectal cancer patients undergoing surgery after long-term or short-term chemoradiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Completeness of mesorectal fascia and specimen quality (specimen integrity after rectal resection) | 4 years
  Specimen quality i.e. integrity of mesorectal fascia and clearance of radial margins are an important factor with impact on local recurrency of rectal cancer. the 3-grade Quirke classification is used to assess completeness of mesorectal fascia: complete, nearly complete and incomplete

SECONDARY OUTCOMES:
Lymph node harvest | 4 years
  The number of lymph nodes harvested may influence patient's prognosis and survival. A minimum number of nodes is required to assess the cancer stage correctly: stage 2 rectal cancer with a less than 12 node harvest has a behaviour of a stage 3 rectal cancer in the medium and long term follow up.
Local recurrence | up to 54-month follow-up (range 6-54 months) with a median follow up respectively 54, 39, 38, 39,5 months for the open TME group, for the laparoscopic TME group, for the robotic TME group and for the TaTME group. Overall median FU = 44 months.
  Local recurrence rate is intended the incidence of pelvic tumor recurrence, especially localized in the presacral area, and anastomotic recurrence
Overal survivals | Overall median follow-up 44 months (FU range 6-54 months), median follow-up per study group: Open TME 54 months, Laparoscopic TME 39 months, Robotic TME 38 months, TaTME 39,5 months.
  short and medium term survivals (Kaplan-Meier estimate)
Cancer specific survival (CSS) | Overall median follow-up 44 months (FU range 6-54 months), median follow-up per study group: Open TME 54 months, Laparoscopic TME 39 months, Robotic TME 38 months, TaTME 39,5 months.
  Cancer-specific survival (CSS) is defined as the duration from the date of diagnosis until death due to rectal cancer other than other causes

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maria Lirici, MD, Principal Investigator — San Giovanni Addolorata Hospital Complex; Saint Camillus International University of Health Sciences
Locations (1):
- San Giovanni Addolorata Hospital Complex, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnajian M, Pettet D 3rd, Kazi E, Foppa C, Bergamaschi R. Quality of total mesorectal excision and depth of circumferential resection margin in rectal cancer: a matched comparison of the first 20 robotic cases. Colorectal Dis. 2014 Aug;16(8):603-9. doi: 10.1111/codi.12634. PMID 24750995
- [Result] Parfitt JR, Driman DK. The total mesorectal excision specimen for rectal cancer: a review of its pathological assessment. J Clin Pathol. 2007 Aug;60(8):849-55. doi: 10.1136/jcp.2006.043802. Epub 2006 Oct 17. PMID 17046842
- [Result] Martellucci J, Bergamini C, Bruscino A, Prosperi P, Tonelli P, Todaro A, Valeri A. Laparoscopic total mesorectal excision for extraperitoneal rectal cancer: long-term results. Int J Colorectal Dis. 2014 Dec;29(12):1493-9. doi: 10.1007/s00384-014-2017-5. Epub 2014 Sep 25. PMID 25248320
- [Result] Havenga K, Grossmann I, DeRuiter M, Wiggers T. Definition of total mesorectal excision, including the perineal phase: technical considerations. Dig Dis. 2007;25(1):44-50. doi: 10.1159/000099169. PMID 17384507
- [Result] Pai A, Marecik SJ, Park JJ, Melich G, Sulo S, Prasad LM. Oncologic and Clinicopathologic Outcomes of Robot-Assisted Total Mesorectal Excision for Rectal Cancer. Dis Colon Rectum. 2015 Jul;58(7):659-67. doi: 10.1097/DCR.0000000000000385. PMID 26200680
- [Result] Heald RJ, Husband EM, Ryall RD. The mesorectum in rectal cancer surgery--the clue to pelvic recurrence? Br J Surg. 1982 Oct;69(10):613-6. doi: 10.1002/bjs.1800691019. PMID 6751457
- [Result] Lacy AM, Tasende MM, Delgado S, Fernandez-Hevia M, Jimenez M, De Lacy B, Castells A, Bravo R, Wexner SD, Heald RJ. Transanal Total Mesorectal Excision for Rectal Cancer: Outcomes after 140 Patients. J Am Coll Surg. 2015 Aug;221(2):415-23. doi: 10.1016/j.jamcollsurg.2015.03.046. Epub 2015 Mar 30. PMID 26206640
- [Result] de Lacy AM, Rattner DW, Adelsdorfer C, Tasende MM, Fernandez M, Delgado S, Sylla P, Martinez-Palli G. Transanal natural orifice transluminal endoscopic surgery (NOTES) rectal resection: "down-to-up" total mesorectal excision (TME)--short-term outcomes in the first 20 cases. Surg Endosc. 2013 Sep;27(9):3165-72. doi: 10.1007/s00464-013-2872-0. Epub 2013 Mar 22. PMID 23519489
- [Result] Velthuis S, Nieuwenhuis DH, Ruijter TE, Cuesta MA, Bonjer HJ, Sietses C. Transanal versus traditional laparoscopic total mesorectal excision for rectal carcinoma. Surg Endosc. 2014 Dec;28(12):3494-9. doi: 10.1007/s00464-014-3636-1. Epub 2014 Jun 28. PMID 24972923
- [Result] van der Pas MH, Haglind E, Cuesta MA, Furst A, Lacy AM, Hop WC, Bonjer HJ; COlorectal cancer Laparoscopic or Open Resection II (COLOR II) Study Group. Laparoscopic versus open surgery for rectal cancer (COLOR II): short-term outcomes of a randomised, phase 3 trial. Lancet Oncol. 2013 Mar;14(3):210-8. doi: 10.1016/S1470-2045(13)70016-0. Epub 2013 Feb 6. PMID 23395398
- [Result] Lino-Silva LS, Garcia-Gomez MA, Aguilar-Romero JM, Dominguez-Rodriguez JA, Salcedo-Hernandez RA, Loaeza-Belmont R, Ruiz-Garcia EB, Herrera-Gomez A. Mesorectal pathologic assessment in two grades predicts accurately recurrence, positive circumferential margin, and correlates with survival. J Surg Oncol. 2015 Dec;112(8):900-6. doi: 10.1002/jso.24076. Epub 2015 Oct 21. PMID 26487289